CLINICAL TRIAL: NCT04269876
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effects of a Specialized Pro-Resolving Mediator Formulation on Inflammation in Individuals Who Are Overweight to Mildly Obese and Otherwise Generally Healthy
Brief Title: A Study to Evaluate the Effects of a Marine Lipid Oil Concentrate Formulation on Inflammation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CL103
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-07

CONDITIONS: Inflammation; Inflammatory Response
MeSH Terms: conditions — Inflammation | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marine Lipid Oil concentrate (Experimental): Dietary Supplement: Marine Lipid oil concentrate softgel and dietary supplement capsules
  Interventions: Dietary Supplement: Marine Lipid Oil Concentrate; Dietary Supplement: Dietary Supplement
- Placebo (Placebo Comparator): Placebo softgels with Placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Marine Lipid Oil Concentrate — Marine Lipid Oil Concentrate softgels
  Arms: Marine Lipid Oil concentrate
Dietary Supplement: Dietary Supplement — Dietary Supplement capsules
  Arms: Marine Lipid Oil concentrate
Dietary Supplement: Placebo — Placebo softgels
  Arms: Placebo
Dietary Supplement: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of a Marine Lipid Oil Concentrate formulation on inflammatory biomarkers and overall well-being in male and female subjects who are overweight to mildly obese, but otherwise generally healthy.

DETAILED DESCRIPTION:
This is a double-blind randomized, placebo-controlled study to evaluate the effects of a Marine Lipid Oil Concentrate formulation on inflammation.. Each subject will receive a specific dose of the study product (A) to be taken once daily with a specific dose of the study product (B) to be taken once daily for a total of 60 days.

Participants will receive questionnaires, assessments, blood tests, vital signs and a body composition analysis.

The primary objective is the assessment of the change in the blood levels of hs-CRP in response to the Marine Lipid Oil Concentrate formulation relative to screening/baseline compared to placebo.

The secondary objective is the assessment of the change in the in response to the Marine Lipid Oil Concentrate formulation relative to screening/baseline compared to placebo for Interleukin-6 (IL-6), Tumor necrosis factor (TNF-alpha), Erythrocyte Sedimentation Rate (ESR), Fibrinogen Activity, B-type natriuretic peptide (BNP), Ferritin, Blood lipid levels (Total Cholesterol, High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), Triglycerides), Short Form-36 (SF-36) Health Survey scores and the Medical Symptoms Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 35-75 years of age
2. A BMI of 23-34.9
3. hs-CRP level of 1-7.5 mg/L
4. Generally healthy and having no significant difficulty with digestion or absorption of food
5. Has been generally weight stable for the past six months (+/- 6 lbs.)
6. Willing and able to give written informed consent
7. Clearly understands the procedures and study requirements
8. Willing and able to comply with all study procedures, including following the recommendations to maintain their usual diet and regular activity, as per protocol
9. Able to communicate, including reading, in English
10. Have not taken any nutritional supplements that may contain any of the components of the study product for a minimum of 14 days before Screening/baseline

Exclusion Criteria:

1. Having smoked any cigarette, electronic cigarette, cigar, pipe, or used a recreational drug as well as any product containing cannabidiol (CBD) and tetrahydrocannabinol in the past 30 days.
2. Donated blood within 30 days before Screening/baseline
3. Inability to provide a venous blood sample
4. Participation in another study within 30 days before Screening/baseline
5. Being pregnant or planning on becoming pregnant during study participation; or breast feeding
6. History of allergy or sensitivity to any component of the study products
7. Currently taking a lipid lowering medication or dietary supplement
8. Currently taking a medication or dietary supplement specifically for pain or inflammation including curcumin and unwilling to washout (i.e., stop taking) for 14 days before Screening/baseline
9. Currently taking or having taken a fish oil, krill oil, omega-3 supplement and omega-3 prescription drugs within the past 3 months before Screening/baseline
10. Currently taking or having taken pain medications or anti-inflammatory medication(s) (e.g., aspirin, NSAIDs, Cyclooxygenase-2 (COX-2) inhibitors, and corticosteroids) within 14 days before Screening/baseline or in the judgment of the Study Investigator/Sub-I would not preclude participation in the study
11. Having been diagnosed, received medical treatment, or taking medication daily for the following medical condition(s):

    * Acute or chronic inflammatory or autoimmune disease (including rheumatoid arthritis, system lupus erythematosus, ankylosing spondylitis, Sjögren's syndrome, polymyalgia rheumatica, inflammatory bowel disease, and psoriatic arthritis)
12. Presence of active or recurring clinically significant conditions as follows:

    * Diabetes mellitus or other endocrine disease
    * Acute infection
    * Active periodontal disease
    * Cardiovascular disease including heart and blood vessel disease, arrhythmia, heart attack, stroke, or heart valve problem
    * Gastrointestinal disease including gallbladder problems, gallstones, or biliary tract obstruction
    * Thyroid disease (unless on a stable dose of medication for 3 months before screening and unlikely to change medication or dose during the study)
    * Hypertension (unless on a stable dose of medication for 3 months screening and unlikely to change medication or dose during the study)
    * Neurologic condition/disease
    * Cancer (unless skin cancer other than melanoma which has been treated > 3 years before Screening/baseline)
    * Liver, pancreatic, and kidney disease
    * Pulmonary disease
    * Blood coagulation disorder or other hematologic disease
    * Other condition or medication use that would preclude participation in the study in the judgment of the Investigator/Sub-I
13. Currently taking any medications or treatment for a psychiatric disorder (bipolar disorder,manic disorder, schizophrenia, apathetic [inherited] disorder), that include antidepressant drugs, including selective serotonin reuptake inhibitors (SSRIs), tricyclic and atypical antidepressants; benzodiazepines; central nervous system (CNS) depressants, dextromethorphan, meperidine, monoamine oxidase inhibitors (MAOIs); pentazocine, phenothiazines, and tramadol. These may preclude participation in the study dependent on the judgment of the Investigator/Sub-I.
14. Currently taking or having taken within the 30 days before Screening/baseline any hormone replacement therapy (including dehydroepiandrosterone (DHEA), estrogen, progesterone, or testosterone; except those utilized as a method of birth control and which have been taken for > 3 months, with no anticipated change for the duration of the study)
15. Having had a surgical procedure or having an internal medical device which, in the judgment of the Study Investigator/Sub-I, would preclude participation in the study
16. Having abnormal screening laboratory test values including bilirubin > 2.5 x upper limit of normal (ULN), aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine transaminase (ALT)/serum glutamic-pyruvic transaminase (SGPT) > 2.5 x ULN, serum creatinine > 1.5 mg/dL, blood glucose < 85 mg/dL or > 110 mg/dL, hs-CRP < 1.0 mg/L or > 5 mg/L, or other lab test result(s) that would preclude study participation in the judgement of the Study Investigator/Sub-I
17. Having blood pressure readings at Screening/baseline > 140 systolic or > 90 diastolic on two consecutive readings unless permitted to proceed to the next visit in the judgment of the Study Investigator/Sub-I
18. Currently consumes more than 7 standard alcoholic drinks per week for women and 14 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
19. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges, and tangelos
20. History of known or suspected substance abuse (e.g., alcohol, opiates, benzodiazepines or amphetamines).
21. Having any other circumstance that precludes study participation in the judgment of the Study Investigator/Sub-I, including use of other nutritional supplements, which will be evaluated on a case-by-case basis.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the mean or median change in high sensitivity C-reactive protein (hs-CRP) relative to baseline | 60 days
  Mean or median change in high sensitivity C-reactive protein (hs-CRP) from baseline to Day 60

SECONDARY OUTCOMES:
Assessment of the mean or median change in Interleukin-6 (IL-6) relative to baseline | 60 days
  Mean or median change in IL-6 from baseline to Day 60
Assessment of the mean or median change in Tumor Necrosis Factor-alpha (TNF-alpha) relative to baseline | 60 days
  Mean or median change in TNF-alpha from baseline to Day 60
Assessment of the mean or median change in Erythrocyte Sedimentation Rate (ESR) relative to baseline | 60 days
  Mean or median change in ESR from baseline to Day 60
Assessment of the mean or median change in Fibrinogen Activity relative to baseline | 60 days
  Mean or median change in Fibrinogen Activity from baseline to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, Ph.D, Principal Investigator — LIfe Extension
Locations (1):
- Lfie Extension Clinical Reseach, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal BB, Gupta SC, Sung B. Curcumin: an orally bioavailable blocker of TNF and other pro-inflammatory biomarkers. Br J Pharmacol. 2013 Aug;169(8):1672-92. doi: 10.1111/bph.12131. PMID 23425071
- [Background] Bassiouny AR, Zaky A, Kandeel KM. Alteration of AP-endonuclease1 expression in curcumin-treated fibrotic rats. Ann Hepatol. 2011 Oct-Dec;10(4):516-30. PMID 21911894
- [Background] Buhrmann C, Mobasheri A, Busch F, Aldinger C, Stahlmann R, Montaseri A, Shakibaei M. Curcumin modulates nuclear factor kappaB (NF-kappaB)-mediated inflammation in human tenocytes in vitro: role of the phosphatidylinositol 3-kinase/Akt pathway. J Biol Chem. 2011 Aug 12;286(32):28556-66. doi: 10.1074/jbc.M111.256180. Epub 2011 Jun 13. PMID 21669872
- [Background] Campbell, M., Berrones, A., Krishnakumar, I. M., Charnigo, R. J., Westgate, P. M., & Fleenor, B. S. (2017). Responsiveness to curcumin intervention is associated with reduced aortic stiffness in young, obese men with higher initial stiffness. J Funct Foods, 29, 154-160.
- [Background] Campbell MS, Ouyang A, I M K, Charnigo RJ, Westgate PM, Fleenor BS. Influence of enhanced bioavailable curcumin on obesity-associated cardiovascular disease risk factors and arterial function: A double-blinded, randomized, controlled trial. Nutrition. 2019 Jun;62:135-139. doi: 10.1016/j.nut.2019.01.002. Epub 2019 Jan 11. PMID 30889454
- [Background] Chainani-Wu N, Madden E, Lozada-Nur F, Silverman S Jr. High-dose curcuminoids are efficacious in the reduction in symptoms and signs of oral lichen planus. J Am Acad Dermatol. 2012 May;66(5):752-60. doi: 10.1016/j.jaad.2011.04.022. Epub 2011 Sep 9. PMID 21907450
- [Background] Chen FY, Zhou J, Guo N, Ma WG, Huang X, Wang H, Yuan ZY. Curcumin retunes cholesterol transport homeostasis and inflammation response in M1 macrophage to prevent atherosclerosis. Biochem Biophys Res Commun. 2015 Nov 27;467(4):872-8. doi: 10.1016/j.bbrc.2015.10.051. Epub 2015 Oct 19. PMID 26471308
- [Background] Dallal, G (2017). Randomization.com. Retrieved from http://www.randomization.com
- [Background] Doyle R, Sadlier DM, Godson C. Pro-resolving lipid mediators: Agents of anti-ageing? Semin Immunol. 2018 Dec;40:36-48. doi: 10.1016/j.smim.2018.09.002. Epub 2018 Oct 4. PMID 30293857
- [Background] Fiala M, Terrando N, Dalli J. Specialized Pro-Resolving Mediators from Omega-3 Fatty Acids Improve Amyloid-beta Phagocytosis and Regulate Inflammation in Patients with Minor Cognitive Impairment. J Alzheimers Dis. 2016;49(4):1191. doi: 10.3233/JAD-159008. No abstract available. PMID 26756328
- [Background] Hewlings SJ, Kalman DS. Curcumin: A Review of Its Effects on Human Health. Foods. 2017 Oct 22;6(10):92. doi: 10.3390/foods6100092. PMID 29065496
- [Background] Krishnakumar, I, Abhilash, M., Gopakumar, G.,et al. Improved blood-brain-barrier permeability and tissue distribution following the oral administration of a food-grade formulation of curcumin with fenugreek fibre. J. Funct Foods, 14, 215-225
- [Background] T Krishnareddy N, Thomas JV, Nair SS, N Mulakal J, Maliakel BP, Krishnakumar IM. A Novel Curcumin-Galactomannoside Complex Delivery System Improves Hepatic Function Markers in Chronic Alcoholics: A Double-Blinded, randomized, Placebo-Controlled Study. Biomed Res Int. 2018 Sep 23;2018:9159281. doi: 10.1155/2018/9159281. eCollection 2018. PMID 30345312
- [Background] Kumar, D., Jacob, D., Subash. P. et al. (2016). Enhanced bioavailability and relative distribution of free (unconjugated) curcuminoids following the oral administration of a food-grade formulation with fenugreek dietary fibre: A randomised double-blind crossover study. J Funt Foods, 22, 578-587
- [Background] Lopez-Vicario C, Rius B, Alcaraz-Quiles J, Garcia-Alonso V, Lopategi A, Titos E, Claria J. Pro-resolving mediators produced from EPA and DHA: Overview of the pathways involved and their mechanisms in metabolic syndrome and related liver diseases. Eur J Pharmacol. 2016 Aug 15;785:133-143. doi: 10.1016/j.ejphar.2015.03.092. Epub 2015 May 15. PMID 25987424
- [Background] Madhu K, Chanda K, Saji MJ. Safety and efficacy of Curcuma longa extract in the treatment of painful knee osteoarthritis: a randomized placebo-controlled trial. Inflammopharmacology. 2013 Apr;21(2):129-36. doi: 10.1007/s10787-012-0163-3. Epub 2012 Dec 16. PMID 23242572
- [Background] Mehra MR, Lavie CJ, Ventura HO, Milani RV. Fish oils produce anti-inflammatory effects and improve body weight in severe heart failure. J Heart Lung Transplant. 2006 Jul;25(7):834-8. doi: 10.1016/j.healun.2006.03.005. Epub 2006 May 24. PMID 16818127
- [Background] Menon VP, Sudheer AR. Antioxidant and anti-inflammatory properties of curcumin. Adv Exp Med Biol. 2007;595:105-25. doi: 10.1007/978-0-387-46401-5_3. PMID 17569207
- [Background] Nathan C, Ding A. Nonresolving inflammation. Cell. 2010 Mar 19;140(6):871-82. doi: 10.1016/j.cell.2010.02.029. PMID 20303877
- [Background] Nordgren TM, Anderson Berry A, Van Ormer M, Zoucha S, Elliott E, Johnson R, McGinn E, Cave C, Rilett K, Weishaar K, Maddipati SS, Appeah H, Hanson C. Omega-3 Fatty Acid Supplementation, Pro-Resolving Mediators, and Clinical Outcomes in Maternal-Infant Pairs. Nutrients. 2019 Jan 5;11(1):98. doi: 10.3390/nu11010098. PMID 30621269
- [Background] Norling LV, Ly L, Dalli J. Resolving inflammation by using nutrition therapy: roles for specialized proresolving mediators. Curr Opin Clin Nutr Metab Care. 2017 Mar;20(2):145-152. doi: 10.1097/MCO.0000000000000353. PMID 28002074
- [Background] Norris PC, Skulas-Ray AC, Riley I, Richter CK, Kris-Etherton PM, Jensen GL, Serhan CN, Maddipati KR. Identification of specialized pro-resolving mediator clusters from healthy adults after intravenous low-dose endotoxin and omega-3 supplementation: a methodological validation. Sci Rep. 2018 Dec 21;8(1):18050. doi: 10.1038/s41598-018-36679-4. PMID 30575798
- [Background] Panahi Y, Hosseini MS, Khalili N, Naimi E, Simental-Mendia LE, Majeed M, Sahebkar A. Effects of curcumin on serum cytokine concentrations in subjects with metabolic syndrome: A post-hoc analysis of a randomized controlled trial. Biomed Pharmacother. 2016 Aug;82:578-82. doi: 10.1016/j.biopha.2016.05.037. Epub 2016 Jun 6. PMID 27470399
- [Background] Pandaran Sudheeran S, Jacob D, Natinga Mulakal J, Gopinathan Nair G, Maliakel A, Maliakel B, Kuttan R, Im K. Safety, Tolerance, and Enhanced Efficacy of a Bioavailable Formulation of Curcumin With Fenugreek Dietary Fiber on Occupational Stress: A Randomized, Double-Blind, Placebo-Controlled Pilot Study. J Clin Psychopharmacol. 2016 Jun;36(3):236-43. doi: 10.1097/JCP.0000000000000508. PMID 27043120
- [Background] Saji S, Asha S, Svenia PJ, Ratheesh M, Sheethal S, Sandya S, Krishnakumar IM. Curcumin-galactomannoside complex inhibits pathogenesis in Ox-LDL-challenged human peripheral blood mononuclear cells. Inflammopharmacology. 2018 Oct;26(5):1273-1282. doi: 10.1007/s10787-018-0474-0. Epub 2018 Apr 9. PMID 29633105
- [Background] Serhan CN. Discovery of specialized pro-resolving mediators marks the dawn of resolution physiology and pharmacology. Mol Aspects Med. 2017 Dec;58:1-11. doi: 10.1016/j.mam.2017.03.001. Epub 2017 Mar 3. PMID 28263773
- [Background] So J, Wu D, Lichtenstein AH, Tai AK, Matthan NR, Maddipati KR, Lamon-Fava S. EPA and DHA differentially modulate monocyte inflammatory response in subjects with chronic inflammation in part via plasma specialized pro-resolving lipid mediators: A randomized, double-blind, crossover study. Atherosclerosis. 2021 Jan;316:90-98. doi: 10.1016/j.atherosclerosis.2020.11.018. Epub 2020 Dec 7. PMID 33303222
- [Background] Spite M, Claria J, Serhan CN. Resolvins, specialized proresolving lipid mediators, and their potential roles in metabolic diseases. Cell Metab. 2014 Jan 7;19(1):21-36. doi: 10.1016/j.cmet.2013.10.006. Epub 2013 Nov 14. PMID 24239568
- [Background] Wongcharoen W, Jai-Aue S, Phrommintikul A, Nawarawong W, Woragidpoonpol S, Tepsuwan T, Sukonthasarn A, Apaijai N, Chattipakorn N. Effects of curcuminoids on frequency of acute myocardial infarction after coronary artery bypass grafting. Am J Cardiol. 2012 Jul 1;110(1):40-4. doi: 10.1016/j.amjcard.2012.02.043. Epub 2012 Apr 3. PMID 22481014
- [Background] Yu Y, Shen Q, Lai Y, Park SY, Ou X, Lin D, Jin M, Zhang W. Anti-inflammatory Effects of Curcumin in Microglial Cells. Front Pharmacol. 2018 Apr 20;9:386. doi: 10.3389/fphar.2018.00386. eCollection 2018. PMID 29731715